CLINICAL TRIAL: NCT06652295
Title: The Effectiveness of Self-Physiotherapy in the Management of Lymphedema Following Breast Cancer Treatment
Brief Title: Effectiveness of Self-Physiotherapy in the Management of Lymphedema
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Sukriye Cansu Gultekin, Principle Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DEU-FTR-SCG-01
Record Dates: First submitted 2024-10-09; First posted 2024-10-22 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer; Lymphedema; Self Care; Quality of Healthcare; Self Management
Keywords: Breast cancer; Upper extremity lymphedema; Complex Decongestive Physiotherapy; Self Management; Health-Related Quality of Life
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: An independent assessor who is unaware of the group of participants going to perform all evaluations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention/Treatment (Active Comparator): This group was enrolled in a complex decongestive physiotherapy programme administered by a physiotherapist five days a week for three weeks.
  Interventions: Other: Complex decongestive physiotherapy (CDP)
- Self-administered Group (Other): This group was enrolled in a self-administered complex decongestive physiotherapy programme five days a week for three weeks.
  Interventions: Other: Self-administered Complex Decongestive Physiotherapy (CDP)

INTERVENTIONS:
Other: Complex decongestive physiotherapy (CDP) — CDP consists of patient education, manual lymph drainage, short traction bandaging, skin/nail care and exercise. The applications of all modalities of the CDP programme were performed by the physiotherapist.
  Arms: Intervention/Treatment
Other: Self-administered Complex Decongestive Physiotherapy (CDP) — The self-administered CDP programme consisted of patient education, self-manual lymph drainage, self-short traction bandage application, self-skin/nail care and exercise. Participants were given one session of patient education before the self-administered CDP programme and patients were given practical information about all applications. Additionally, each component of the self-administered CDP programme was presented to the participants with a patient booklet and a video prepared by the researchers. Patients in the self-CDP group were followed up once a week with a patient follow-up diary.
  Arms: Self-administered Group

SUMMARY:
Breast cancer-related lymphedema is a chronic condition adversely affecting physical, social, psychological and emotional well-being. The complex decongestive physiotherapy (CDP) programme is considered the gold standard in the management of lymphedema. The most important barriers affecting patient participation in the CDP programme are the lack of trained health personnel and the difficulty for patients to access treatment (peripheral location or financial difficulties). Therefore, self-administration of the CDP programme may contribute to the development of self-care strategies and the reduction of treatment costs.

DETAILED DESCRIPTION:
Breast cancer (BC) is the most common type of cancer in women according to the GLOBOCAN cancer data. The advancements in BC screening, diagnosis and treatment have increased the 5-year survival rate to more than 90%. On the other hand, the chronic disease process and side effects of treatment in BC survivors have been reported to lead to significant morbidities. Breast cancer-related lymphedema (BCRL) is reported as one of the most common morbidities leading to impaired upper extremity functionality and decreased quality of life. Lymphedema is a chronic condition characterized by abnormal accumulation of protein-rich fluid in the interstitial space due to insufficient lymphatic drainage. Complex decongestive physiotherapy (CDP) (patient education, manual lymph drainage, compression, exercise, skin care) programme is considered the gold standard modality in the management of lymphedema. On the other hand, the CDP programme is time-consuming, the high cost of health expenditures and the insufficient number of health personnel with expertise in the field are the major barriers for BCRL patients to participate in the CDP programme. Additionally, some of the patients have difficulties in reaching the treatment due to their peripheral locations. Moreover, considering the chronic nature of lymphedema, patients usually require several CDP application for the management of lymphedema throughout their life. Therefore, the development of self-management programme which are transferable across regional and economic boundaries might emerge as an important approach to reduce healthcare costs and improve long-term outcomes in lymphedema management. Most studies of self-management in lymphedema focus on patient education and for using compression garments. On the other hand, recent findings have suggested the most effective approach to lymphedema management is to incorporate all components of the CDP programme as a multimodal approach. Therefore, this study aims to investigate the feasibility of the CDP protocol as a self-management treatment option by BCRL patients. Self-administered CDP protocol may be a practice that enables the patient to adopt self-care activities, reducing treatment costs and physiotherapist workload. The primary aim of the study was to compare the effectiveness of self-management and physiotherapist-administered CDP on lymphedema severity in patients with BCRL. The secondary aim was to compare the efficacy of self-management and physiotherapist-administered CDP on disease-related clinical outcomes in patients with BCRL.

The study is a single-blind randomized controlled study with pre-test post-test design. The study consisted of a total of 50 BCRL patients, 25 in the standard treatment (CDP administered by a physiotherapist) group and 25 in the self-administered CPD group.

Participants were randomly assigned to one of two possible experimental conditions: (1) a physiotherapist-administered CDP programme or (2) a self-administered CDP programme. The CDP programme consisted of patient education, manual lymph drainage, short traction bandaging and remedial exercises. Before the CDP programme, the participants were provided one session of patient education and the patients were informed about all applications. Each component of the self-CDP programme was presented to the participants with a lymphedema patient booklet and a video prepared by the researchers. Both experimental groups enrolled in the study for five days a week for three weeks. Patients in the Self-CDP group was followed up once a week with a patient follow-up diary. A blinded physiotherapist performed all pre- and post-treatment assessments. Breast cancer (BC) is the most common type of cancer in women according to the GLOBOCAN cancer data. The advancements in BC screening, diagnosis and treatment have increased the 5-year survival rate to more than 90%. On the other hand, the chronic disease process and side effects of treatment in BC survivors have been reported to lead to significant morbidities. Breast cancer-related lymphedema (BCRL) is reported as one of the most common morbidities leading to impaired upper extremity functionality and decreased quality of life. Lymphedema is a chronic condition characterized by abnormal accumulation of protein-rich fluid in the interstitial space due to insufficient lymphatic drainage. Complex decongestive physiotherapy (CDP) (patient education, manual lymph drainage, compression, exercise, skin care) programme is considered the gold standard modality in the management of lymphedema. On the other hand, the CDP programme is time-consuming, the high cost of health expenditures and the insufficient number of health personnel with expertise in the field are the major barriers for BCRL patients to participate in the CDP programme. Additionally, some of the patients have difficulties in reaching the treatment due to their peripheral locations. Moreover, considering the chronic nature of lymphedema, patients usually require several CDP application for the management of lymphedema throughout their life. Therefore, the development of self-management programme which are transferable across regional and economic boundaries might emerge as an important approach to reduce healthcare costs and improve long-term outcomes in lymphedema management. Most studies of self-management in lymphedema focus on patient education and for using compression garments. On the other hand, recent findings have suggested the most effective approach to lymphedema management is to incorporate all components of the CDP programme as a multimodal approach. Therefore, this study aims to investigate the feasibility of the CDP protocol as a self-management treatment option by BCRL patients. Self-administered CDP protocol may be a practice that enables the patient to adopt self-care activities, reducing treatment costs and physiotherapist workload. The primary aim of the study was to compare the effectiveness of self-management and physiotherapist-administered CDP on lymphedema severity in patients with BCRL. The secondary aim was to compare the efficacy of self-management and physiotherapist-administered CDP on disease-related clinical outcomes in patients with BCRL.

The study is a single-blind randomized controlled study with pre-test post-test design. The study consisted of a total of 50 BCRL patients, 25 in the standard treatment (CDP administered by a physiotherapist) group and 25 in the self-administered CPD group.

Participants were randomly assigned to one of two possible experimental conditions: (1) a physiotherapist-administered CDP programme or (2) a self-administered CDP programme. The CDP programme consisted of patient education, manual lymph drainage, short traction bandaging and remedial exercises. Before the CDP programme, the participants were provided one session of patient education and the patients were informed about all applications. Each component of the self-CDP programme was presented to the participants with a lymphedema patient booklet and a video prepared by the researchers. Both experimental groups enrolled in the study for five days a week for three weeks. Patients in the Self-CDP group was followed up once a week with a patient follow-up diary. A blinded physiotherapist performed all pre- and post-treatment assessments.Participants will be recalled after 3 months for re-assessment of lymphoedema severity and symptoms.

ELIGIBILITY:
* Being 18 years of age or older
* Having stage 1-3 lymphedema according to the International Society of Lymphology (ISL) classification
* Having a diagnosis of unilateral breast cancer-related lymphedema (Doppler, lymphoscintigraphy, and computed tomography were preferred to confirm the diagnosis of lymphedema based on a comprehensive medical assessment and condition of the patient)
* No evidence/suspicion of cancer recurrence after completion of adjuvant local and systemic therapies for at least 12 months
* Not having received a complex decongestive physiotherapy programme in the last 6 months
* Volunteer to participate in the study Able to read and understand Turkish.

Exclusion Criteria:

* Inability to understand the questionnaires and refusal to participate
* History of congenital lymphedema or bilateral upper extremity lymphedema or malignant lymphedema
* Presence of neurological or mental illness or axillary web syndrome, major organ failure, or/ iatrogenic disease that may adversely affect the severity of lymphedema (such as using steroids, nonsteroidal anti-inflammatory drugs, and calcium channel blockers)
* Presence of conditions contraindicated for complex decongestive physiotherapy (active infection, deep vein thrombosis/thrombophlebitis, cardiac oedema, pulmonary disease, peripheral arterial disease, any skin disease such as scleroderma, allergic reactions to treatment).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-01-25 (Estimated)

PRIMARY OUTCOMES:
Edema severity | Change from oedema severity baseline at 3 weeks (end of treatment) to 3 months (follow-up sessions)
  The severity of lymphedema was evaluated by circumferential measurement. The circumference of both limbs was measured starting from the nail base of the third finger to the proximal part at 5 cm intervals. The difference between both arms was recorded in cm. The severity of edema was evaluated according to the criteria determined by the American Physical Therapy Association. According to these criteria, a difference of less than 3 cm between both limbs was recorded as mild severity, 3-5 cm as moderate severity, and greater than 5 cm as severe lymphedema.
Symptom Assessment | Change from baseline symptoms at 3 weeks (end of treatment) to 1 month and 3 months (follow-up sessions)
  A numerical scale from 0 to 10 was used for symptom assessment (severity of pain, swelling, feeling of heaviness, increased temperature, feeling of tightness, fatigue, numbness and tingling). A numerical scale from 0 to 10 was used to report severity. 0 indicates no complaints; 10 indicates intolerable complaints.

SECONDARY OUTCOMES:
Range of Motion | Change from baseline upper extremity range of motion at 3 weeks (end of treatment)
  The upper extremity range of motion of the participants was evaluated as bilateral. Upper extremity shoulder flexion, abduction, internal rotation, external rotation, elbow flexion, extension, wrist flexion and extension were measured with a standard goniometer using standard measurement procedures.
Hand grip strength | Change from baseline hand grip strength at 3 weeks (end of treatment)
  Hand grip strength was measured with a hydraulic hand dynamometer (Jamar, Sammons Preston Rolyan, Chicago, USA). Patients were instructed to perform a maximum isometric contraction. The test was repeated within 30 seconds and the highest value of the three tests was used for analysis.
Assessment of Physical Activity Level | Change from baseline physical activity level at 3 weeks (end of treatment)
  The International Physical Activity Questionnaires (IPAQ) - short form was used to inquire about the physical activity levels of the participants. This questionnaire consists of seven questions asking participants to remember the last week's physical activity. The IPAQ-short form inquiries about the number of days and amount of the spent walking, sitting or participating in moderate (e.g., bicycling at a regular pace) and vigorous-intensity activities (e.g., fast bicycling, digging) and reports the frequency and duration of these activity. Higher scores indicate higher levels of physical activity.
Patient Benefit Index | Change from baseline patient benefit index score at 3 weeks (end of treatment)
  The benefit that participants received from treatment was measured using the Patient Benefit Index - Lymphedema. This questionnaire is a measure of the importance of treatment goals to the patient and the degree of benefit from treatment. The questionnaire is divided into two distinct sections: "Treatment Goals" and "Treatment Benefits". Each section contains 23 questions, for a total of 46 questions. The answers are scored on a scale of 0 to 4, with the following descriptors being used 'Doesn't affect me', 'Doesn't affect me at all', 'A little', 'Moderately', 'A lot' and 'Very much'. Higher scores indicate more perceived benefit from the treatment.
Health Related Quality of Life Assesment | Change from baseline symptoms at 3 weeks (end of treatment)
  The Upper Limb Lymphedema 27 (ULL-27) questionnaire was used to assess the impact of arm function on quality of life in patients with lymphedema. The scale consists of 27 questions with physical, psychological and social dimensions. A 5-point Likert scale (1=strongly disagree, 5=strongly agree) is used. The first 15 questions assess the physical dimension (minimum 15 and maximum 75 points), questions between 16 and 22 assess the social dimension (minimum 7 and maximum 35 points) and questions between 23 and 27 assess the social dimension (minimum 5 points). The total score of the 27 questions is calculated for the overall score. The lowest score is 27 and the highest is 135. A high score on the scale indicates a negative impact on the quality of life of the patient.
Upper Extremity Disability Level | Change from baseline upper extremity disability level at 3 weeks (end of treatment)
  DASH will be used to measure the level of upper extremity-related disability. The questionnaire consists of 30 items divided into 2 subcategories: disability/symptom scores and work module scores. Each item is rated on a 5-point Likert scale (1 to 5). The total score ranges from 0 to 100, with higher scores indicating greater upper extremity-related disability.
Fatigue | Change from baseline symptoms at 3 weeks (end of treatment)
  The Checklist Individual Strength (CIS) will utilized for assessing fatigue levels. The CIS is a valid and reliable tool to evaluate fatigue in cancer patients. The questionnaire consists of 20 items and four dimensions: the subjective feeling of fatigue (eight items), motivation (four items), physical activity (three items), and concentration (five items). A higher score on the CIS indicates a greater degree of fatigue, decreased motivation, reduced physical activity, and concentration difficulties.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and the need to protect sensitive personal health information. Additionally, the lack of a comprehensive data-sharing agreement among collaborators may hinder the ability to share data responsibly. At this stage, there is also no formal infrastructure in place to manage and safeguard shared data effectively.